CLINICAL TRIAL: NCT00235755
Title: Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group Phase 3 Study - Determine Efficacy and Safety of Two Doses of Retigabine (900 Mg/Day and 600 Mg/Day) Used as Adjunctive Therapy in Refractory Epilepsy Patients With Partial-Onset Seizures
Brief Title: Retigabine Efficacy and Safety Trial for Partial Onset Refractory Seizures in Epilepsy
Acronym: RESTORE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VRX-RET-E22-302
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Results first posted 2011-11-07 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Seizures
Keywords: Partial Seizures; Complex Partial Seizures; Epilepsy; Potassium Channels; Anticonvulsant
MeSH Terms: conditions — Seizures; Epilepsy | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Retigabine 600 mg (Experimental)
  Interventions: Drug: Retigabine
- Retigabine 900 mg (Experimental)
  Interventions: Drug: Retigabine

INTERVENTIONS:
Drug: Retigabine — Oral tablet. The starting daily dose will be 300 mg/day administered orally in three equally divided doses. This dosage will be increased by 150 mg/day (50 mg/dose) at 1-week intervals (titration phase). At the beginning of Week 3, patients will enter a 12 week maintenance phase.
  Other Names: GKE-841; D-23129
  Arms: Retigabine 600 mg
Drug: Retigabine — Oral tablet. The starting daily dose will be 300 mg/day administered orally in three equally divided doses. This dosage will be increased by 150 mg/day (50 mg/dose) at 1-week intervals (titration phase). At the beginning of Week 5, patients will enter a 12 week maintenance phase.
  Other Names: GKE-841; D-23129
  Arms: Retigabine 900 mg
Drug: Placebo — Oral tablet.
  Arms: Placebo

SUMMARY:
This Phase 3 study is being conducted to evaluate the efficacy and safety of retigabine dosed at 900 mg/day and 600 mg/day, in three equally divided doses, compared with placebo in patients with epilepsy who are receiving up to three established antiepileptic drugs (AEDs).

DETAILED DESCRIPTION:
This Phase 3 study is being conducted in Europe, Israel, Australia, and South Africa to evaluate the efficacy and safety of retigabine dosed at 900 mg/day and 600 mg/day, in three equally divided doses, compared with placebo in patients with epilepsy who are receiving up to three established antiepileptic drugs (AEDs). The primary objective is to demonstrate a superior change in total partial seizure frequency for four weeks from baseline to the double-blind period. The proportion of responders (greater than or equal to 50% reduction in seizure frequency for four weeks from baseline to the double-blind period) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory epilepsy with simple or complex partial onset seizures with or without secondary generalization
* 28-day partial seizure frequency rate of four or more partial seizures over the 8-week baseline phase
* Currently treated with up to three established AEDs
* Vagal Nerve Stimulator may be included

Exclusion Criteria:

* Existing medical or psychiatric condition which could affect patient's health or compromise ability to participate in the study
* Clinically significant abnormalities on physical exam, vital signs, ECG, or liver function tests
* Impaired renal function (creatinine clearance less than 50 mL/minute)
* Evidence of progressive central nervous disease, lesion, or encephalopathy
* History of primary generalized seizures
* History of clustering or flurries or status epilepticus within 12 months of study entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2005-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (70):
- United States (2):
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Neurological Clinic-Texas, Dallas, Texas
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - North Coast Neurology Centre, Maroochydore, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Austin & Repatriation Medical Centre, West Heidelberg, Victoria
- Belgium (4):
  - A. Z. Middelheim -- Department of Neurology, Antwerp
  - AZ Sint-Jan, Bruges
  - Universitaire Ziekenhuizen Gasthuisberg -- Department Neurology, Leuven
  - Centre Neurologique William Lennox, Ottignies
- France (4):
  - Hopital Neurologique Pierre Wertheimer, Lyon, Lyonnais
  - CHU Pontchaillou, Rennes
  - Hopital Civil de Strasbourg, Strasbourg
  - Centre Medical de La Teppe, Tain-l'Hermitage
- Germany (7):
  - University of Bonn -- Department for Epileptplogy, Bonn
  - Zentrum Epilepsie Erlangen (ZEE) der Universitaet Erlangen, Erlangen
  - Georg-August-Universitaet Goettingen, Göttingen
  - Universitaetsklinik Mainz Neurologische Klinik, Mainz
  - Universitaet Giessen / Marburg Neurologie, Marburg
  - Theatinerstrasse 44, Munich
  - Universitaetsklinikum Ulm, Ulm
- Hungary (2):
  - Natl. Inst. of Psychiatry and Neurology, Budapest
  - Orszagos Idegsebeszeti Tudomanyos Intezet, Budapest
- Israel (8):
  - Barzilai Medical Center, Ashkelon
  - Assaf Harofeh Medical Center, Beer Yaakov
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Western Galilee Hospital, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Poland (7):
  - Specjalistyczna Przychodnia Lekarska Medikard, Padlewskiego 4, Plock
  - NZOZ Przychodnia Internistyczno - Stomatologiczna "Kendron", Bialystok
  - Wojewodzki Szpital Specjalistyczny im.Mikolaja Kopernika, Gdansk
  - Katedra i Klinika Neurologii Slaskiej Akademii Medycznej, Katowice
  - WSS im.Kardynala S. Wyszynskiego, Lublin
  - Instytut Psychiatrii i Neurologii II Oddzial Neurologii, Warsaw
  - Prywatna Wielospecjalistyczna Lecznica Medyczna "Zycie", Warsaw
- Russia (6):
  - Interregional Clinical Diagnostic Centre, Kazan'
  - City Hospital # 1, Moscow
  - Clinic of Nervous Diseases of Sechenov's Moscow Med. Academy, Moscow
  - District Antiepileptic Centre City Clinical Hospital # 71, Moscow
  - Military Medical Academy n.a. S.M.Kirov, Saint Petersburg
  - St.Petersburg State Medical University n.a. I.P.Pavlov, Saint Petersburg
- South Africa (9):
  - Triple M Research, Port Elizabeth, East Cape
  - University of the Free State, Bloemfontein, Gauteng
  - Wilgers MR & Medical Centre, Pretoria, Gauteng
  - Sunninghill & Kopano Clinical Trials, Sunninghill, Gauteng
  - Johannesburg Hospital, Johannesburg, Gauten
  - Inkosi Albert Luthuli Central Hospital, Durban, KwaZulu-Natal
  - Carl Bremer Hospital, Belville, West Cape
  - Groote Schuur Hospital, Cape Town, Western Cape
  - Panorama Medi-Clinic, Cape Town
- Spain (6):
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital de Cruces, Bilbao
  - Hosp de Donostia, Donostia / San Sebastian
  - Hosp. Virgen de las Nieves, Granada
  - Hospital Ruber Internacional de Madrid, Madrid
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
- Ukraine (5):
  - Psychosomatic Center of Dnepropetr. Regional Clinic, Dnipro
  - Kharkiv State Medical University, Kharkiv
  - Institute of Neurology, Psychiatry and Narcology of AMS, Ukr, Kharkiv
  - Epilepsy Center of Municipal Clinical Psychoneurological Hospital, Kiev
  - Odessa Regional Clinical Hospital, Odesa
- United Kingdom (5):
  - The James Cook University Hospital, Middlesbrough, Mersyd
  - Fylde Coast Hospital, Blackpool
  - Western Infirmary (Epilepsy), Glasgow
  - Walton Centre for Neurology & Neurosurgery, Liverpool
  - Royal London Hospital, London

REFERENCES:
- [Background] Brodie MJ, Lerche H, Gil-Nagel A, Elger C, Hall S, Shin P, Nohria V, Mansbach H; RESTORE 2 Study Group. Efficacy and safety of adjunctive ezogabine (retigabine) in refractory partial epilepsy. Neurology. 2010 Nov 16;75(20):1817-24. doi: 10.1212/WNL.0b013e3181fd6170. Epub 2010 Oct 13. PMID 20944074
- [Background] Tompson DJ, Crean CS. Clinical pharmacokinetics of retigabine/ezogabine. Curr Clin Pharmacol. 2013 Nov;8(4):319-31. doi: 10.2174/15748847113089990053. PMID 23342983
- [Background] Brickel N, Gandhi P, VanLandingham K, Hammond J, DeRossett S. The urinary safety profile and secondary renal effects of retigabine (ezogabine): a first-in-class antiepileptic drug that targets KCNQ (K(v)7) potassium channels. Epilepsia. 2012 Apr;53(4):606-12. doi: 10.1111/j.1528-1167.2012.03441.x. Epub 2012 Mar 16. PMID 22428574
- [Derived] Porter RJ, Burdette DE, Gil-Nagel A, Hall ST, White R, Shaikh S, DeRossett SE. Retigabine as adjunctive therapy in adults with partial-onset seizures: integrated analysis of three pivotal controlled trials. Epilepsy Res. 2012 Aug;101(1-2):103-12. doi: 10.1016/j.eplepsyres.2012.03.010. Epub 2012 Apr 16. PMID 22512894
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: VRX-RET-E22-302 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: VRX-RET-E22-302 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: VRX-RET-E22-302 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: VRX-RET-E22-302 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: VRX-RET-E22-302 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: VRX-RET-E22-302 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: VRX-RET-E22-302 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the Double-blind Phase (Titration plus Maintenance Phases) who elected to continue in the Open-Label Extension Study (OLE-S) entered the Transition Phase, for titration, if on placebo, or to maintain the blind if on retigabine. Participants who did not enter the Titration Phase entered a Taper Phase.
Groups:
- Placebo: Matching placebo tablets of dummy strengths of 50 milligrams (mg) and 100 mg were administered orally thrice a day (TID) during the 4-week Titration Phase. Matching placebo tablets of dummy strengths of 50 mg and 100 mg were administered orally TID during the 12-week Maintenance Phase.
- Retigabine 200 mg TID: Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 200 mg TID during the Titration Phase, during which participants were titrated from 300 mg per day to 600 mg per day with weekly increases in doses of 150 mg per day over the course of 2 to 4 weeks. Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 200 mg TID during the 12-week Maintenance Phase.
- Retigabine 300 mg TID: Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 300 mg TID during the Titration Phase, during which participants were titrated from 300 mg per day to 900 mg per day with weekly increases in doses of 150 mg per day over the course of 2 to 4 weeks. Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 300 mg TID during the 12-week Maintenance Phase.
Period: 4-Week Titration Phase
Arm/Group | Placebo | Retigabine 200 mg TID | Retigabine 300 mg TID
Started | 179 | 181 | 179
Completed | 168 | 162 | 153
Not Completed | 11 | 19 | 26
Not completed — Adverse Event | 6 | 14 | 20
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Protocol Violation | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 3
Not completed — Participant Did Not Receive Study Drug | 0 | 0 | 1
Not completed — Randomization Occurred in Error | 1 | 0 | 0
Not completed — Prolonged QT Interval at Visit 3 | 1 | 0 | 0
Period: 12-Week Maintenance Phase
Arm/Group | Placebo | Retigabine 200 mg TID | Retigabine 300 mg TID
Started | 168 | 162 | 153
Completed | 152 | 135 | 122
Not Completed | 16 | 27 | 31
Not completed — Adverse Event | 8 | 12 | 26
Not completed — Lost to Follow-up | 2 | 3 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0
Not completed — Protocol Violation | 0 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 8 | 3
Not completed — Abnormal Electrocardiogram Test Result | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo - Double Blind (DB) Phase (Titration Plus Maintenance): Matching placebo tablets of dummy strengths of 50 milligrams (mg) and 100 mg were administered orally thrice a day (TID) during the 4-week Titration Phase and the 12-week Maintenance Phase
- Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance): Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 200 mg TID during the Titration Phase, during which participants were titrated from 300 mg per day to 600 mg per day with weekly increases in doses of 150 mg per day over the course of 2 to 4 weeks, followed by a 12-week Maintenance Phase, during which participants were administered 200 mg TID
- Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance): Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 300 mg TID during the Titration Phase, during which participants were titrated from 300 mg per day to 900 mg per day with weekly increases in doses of 150 mg per day over the course of 2 to 4 weeks, followed by a 12-week Maintenance Phase, during which participants were administered 300 mg TID
- Total: Total of all reporting groups
Arm/Group | Placebo - Double Blind (DB) Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance) | Total
Number analyzed (Participants) | 179 | 181 | 178 | 538
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics are summarized for the Safety Population, comprised of all participants who were randomized and received at least one dose of study medication.
  Years | 37.7 (11.75) | 37.5 (12.02) | 37.7 (12.77) | 37.6 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 105 | 85 | 280
  Male | 89 | 76 | 93 | 258
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 169 | 173 | 170 | 512
  African-American (black) | 2 | 2 | 1 | 5
  Asian | 3 | 0 | 2 | 5
  Mixed Race | 5 | 6 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the 28-day Total Partial Seizure (PS) Frequency From Baseline (BL) to the End of the Double-blind (DB) Phase (Titration and Maintenance Phases)
Description: 28-day total PS (PSs [also called focal seizures] are seizures limited to a specific area of the brain) frequency in the BL period = (Number [No.] of total PSs reported in the BL period divided by the No. of days of available total PS data in the BL period) x 28 days. 28-day total PS frequency in the DB period = (No. of total PSs reported in the DB period divided by the No. of days of available total PS data in the DB period) x 28 days. Percent change = ([value in the DB period minus value at BL] divided by the BL value) x 100%. Negative valu es indicate a reduction in seizure frequency.
Time Frame: Baseline (Week -7 through Week 0), DB Phase (Week 1 through Week 16)
Population: Intent-to-Treat Food and Drug Administration (ITT FDA) Population: all randomized participants (P) who received at least 1 dose of study drug. Only participants with post-BL seizure data are included in this analysis.
Measure: Median (Full Range); unit: percent change in seizure frequency
Arm/Group | Placebo - Double Blind (DB) Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 176 | 175 | 179
percent change in seizure frequency | -15.9 [-100 to 1712] | -39.9 [-100 to 226] | -27.9 [-94 to 250]
Statistical Analysis 1: Comparison: Placebo - Double Blind (DB) Phase (Titration Plus Maintenance) vs Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance); Test type: Superiority or Other; p < 0.001, Non-parametric rank ANCOVA — Non-parametric rank analysis of covariance adjusted for baseline 28-seizure frequency and stratified by baseline seizure frequency category and region
Statistical Analysis 2: Comparison: Placebo - Double Blind (DB) Phase (Titration Plus Maintenance) vs Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance); Test type: Superiority or Other; p = 0.007, Non-parametric rank ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Participants Classified as Responders and Non-responders During the Maintenance Phase
Description: Responders were participants with at least a 50% reduction in the 28-day total partial seizure frequency in the Maintenance Phase as compared to the Baseline period.
Time Frame: Week 5 through Week 16
Population: ITT European Medicines Evaluation Agency (EMEA) Population: all randomized participants who had received at least 1 dose of study drug in the Maintenance Phase and had at least 1 seizure measurement (whether or not they had a seizure) recorded in the Maintenance Phase.
Measure: Number; unit: participants
Groups:
- Placebo - DB Phase (Titration Plus Maintenance): Matching placebo tablets of dummy strengths of 50 mg and 100 mg were administered orally TID during the 4-week Titration Phase and the 12 week Maintenance Phase
- Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance: Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 200 mg TID during the Titration Phase, during which participants were titrated from 300 mg per day to 600 mg per day with weekly increases in doses of 150 mg per day over the course of 2 to 4 weeks, followed by a 12-week Maintenance Phase, during which participants were administered 200 mg TID
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance
Number analyzed (Participants) | 164 | 149 | 158
participants
  Responders | 31 | 70 | 61
  Non-responders | 133 | 79 | 97
Statistical Analysis 1: Comparison: Placebo - DB Phase (Titration Plus Maintenance) vs Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance); Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo - DB Phase (Titration Plus Maintenance) vs Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: Number of Participants Who Were Responders and Non-responders During the DB Phase
Description: Responders were participants with at least a 50% reduction in the 28-day total partial seizure frequency in the DB Phase as compared to the Baseline period. Participants without any post-baseline data were considered non-responders.
Time Frame: Week 1 through Week 16
Population: ITT FDA Population
Measure: Number; unit: participants
Groups:
- Placebo - DB Phase (Titration Plus Maintenance): Matching placebo tablets of dummy strengths of 50 mg and 100 mg were administered orally TID during the 4-week Titration Phase and the 12-week Maintenance Phase
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 179 | 181 | 178
participants
  Responders | 31 | 57 | 70
  Non-responders | 148 | 124 | 108

4. Secondary Outcome: Percent Change From Baseline (BL) in the 28-day Total Partial Seizure Frequency During the Maintenance Phase
Description: 28-day total partial seizure frequency in the BL period = (No. of total partial seizures reported in the BL period divided by the No. of days of available total partial seizure data in the BL period) x 28 days. 28-day total partial seizure frequency in the Maintenance Phase = (No. of total partial seizures reported in the Maintenance Phase divided by the No. of days of available total partial seizure data in the same phase) x 28 days. Percent change = (value in the Maintenance Phase minus value at BL divided by the BL value) x 100%. Negative values indicate a reduction in seizure frequency.
Time Frame: Baseline (Week -7 through Week 0), Week 5 through Week 16
Population: ITT EMEA Population
Measure: Median (Full Range); unit: Percent change in seizure frequency
Groups:
- Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance): Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 300 mg TID during the Titration Phase, during which participants were titrated from 300 mg per day to 900 mg per day with weekly increases in doses of 150 mg per day over the course of 2 to 4 weeks followed by a 12-week Maintenance Phase, during which participants were administered 300 mg TID
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 164 | 158 | 149
Percent change in seizure frequency | -17.4 [-100 to 1589] | -35.3 [-100 to 253] | -44.3 [-100 to 714]

5. Secondary Outcome: Number of Participants With a Reduction in the 28-day Total Partial Seizure Frequency From Baseline to the End of DB Phase (Titration and Maintenance Phases) by Indicated Quartile Reduction Categories
Description: Participants who experienced a reduction from Baseline in the 28-day total partial seizure frequency were categorized as having a reduction of 75-100%, 50-<75%, 25-<50%, or <25%, in addition to having no reduction. This quartile cutting was specified in the study protocol. Participants without any post-baseline data are included in the "No reduction" category.
Time Frame: Baseline (Week -7 through Week 0), Week 1 through Week 16
Population: ITT FDA Population
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 179 | 181 | 178
participants
  75% to 100% reduction | 12 | 16 | 27
  50% to <75% reduction | 19 | 41 | 43
  25% to <50% reduction | 39 | 38 | 41
  >0 to <25% reduction | 43 | 38 | 24
  No reduction | 66 | 48 | 43

6. Secondary Outcome: Number of Participants With a Reduction in the 28-day Total Partial Seizure Frequency From Baseline to the DB Phase (Titration and Maintenance Phases) by Indicated Decile Reduction and Increase Categories
Description: Participants who experienced a reduction from Baseline in the 28-day total partial seizure frequency were categorized in decile cutting, i.e., reduction categories of 90-100%, 80-<90%, 70-<80%, 60-<70%, 50-<60%, 40-<50%, 30-<40%, 20-<30%, 10-<20%, >0-<10%, and increase categories of 0-10%, >10-20%, >20-30%, >30% (FDA endpoint). Participants without any post-baseline data were included in the category 0-10% increase category.
Time Frame: Baseline (Week -7 through Week 0), Week 1 through Week 16
Population: ITT FDA Population
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 179 | 181 | 178
participants
  Reduction: 90% to 100% | 3 | 5 | 11
  Reduction: 80% to <90% | 4 | 8 | 14
  Reduction: 70% to <80% | 8 | 11 | 7
  Reduction: 60% to <70% | 7 | 14 | 21
  Reduction: 50% to <60% | 9 | 19 | 17
  Reduction: 40% to <50% | 9 | 13 | 17
  Reduction: 30% to <40% | 15 | 16 | 21
  Reduction: 20% to <30% | 24 | 16 | 9
  Reduction: 10% to <20% | 18 | 18 | 10
  Reduction: >0% to <10% | 16 | 13 | 8
  Increase: 0% to 10% | 20 | 11 | 11
  Increase: >10% to 20% | 13 | 9 | 7
  Increase: >20% to 30% | 8 | 3 | 1
  Increase: >30% | 25 | 25 | 24

7. Secondary Outcome: Number of Participants With the Indicated Reduction From Baseline in the 28-day Total Partial Seizure Frequency During the Maintenance Phase
Description: Participants who experienced a reduction from Baseline in the 28-day total partial seizure frequency were categorized as having a >75%, a 50-75%, or a <50% reduction, in addition to having no reduction (EMEA endpoint).
Time Frame: Baseline (Week -7 through Week 0), Week 5 through Week 16
Population: ITT EMEA Population
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 164 | 158 | 149
participants
  >75% reduction | 11 | 27 | 30
  50% to 75% reduction | 20 | 34 | 40
  >0 to <50% reduction | 83 | 60 | 49
  No reduction | 50 | 37 | 30

8. Secondary Outcome: Number of Participants Who Experienced the Indicated Level of Exacerbation and Reduction in the 28-day Total Partial Seizure Frequency From Baseline During the Maintenance Phase
Description: Participants who experienced an exacerbation from Baseline in the 28-day total partial seizure frequency were categorized as having a 0-25% or a >25% increase (EMEA endpoint). The number of participants experiencing a >0% reduction from Baseline in the 28-day total partial seizure frequency are also presented.
Time Frame: Baseline (Week -7 through Week 0), Week 5 through Week 16
Population: ITT EMEA Population
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 164 | 158 | 149
participants
  0% to 25% increase | 28 | 14 | 11
  >=25% increase | 22 | 23 | 19
  >0% reduction | 114 | 121 | 119

9. Secondary Outcome: Number of Participants Reporting New Seizure Types in the Indicated Categories During the DB Phase (Titration and Maintenance Phases) That Were Not Reported at Baseline
Description: New seizure types included those seizures which were not reported by any participant at Baseline.
Time Frame: Baseline (Week -7 through Week 0), Week 1 through Week 16
Population: ITT FDA Population
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 179 | 181 | 178
participants
  Partial seizures without motor signs | 9 | 8 | 12
  Partial evolving to secondarily generalized | 6 | 5 | 9
  Partial seizures with motor signs | 5 | 6 | 3
  Tonic-clonic seizures | 0 | 0 | 3
  Flurries | 3 | 2 | 1
  Tonic seizures | 3 | 0 | 1
  Complex partial seizures | 1 | 4 | 4
  Unclassified seizures | 0 | 1 | 0

10. Secondary Outcome: Number of Participants Who Were Seizure-free During the DB Phase (Titration and Maintenance Phases)
Description: Participants were considered to be seizure-free if they had not reported any seizures during the DB treatment period (Weeks 1-18). For a participant to be seizure free during the DB Phase, the participant had to be seizure free both Week 7 to Week 18 and Week 1 to Week 6. A participant could be seizure free Week 7 to Week 18 (during the Maintenance Phase), but not seizure free Week 1 to Week 6. Hence, there are fewer participants being reported as seizure free from Week 1 to Week 18 than from Week 7 to Week 18.
Time Frame: Week 1 through Week 16
Population: ITT FDA Population. Only participants with post-baseline seizure data were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 176 | 179 | 175
participants
  Seizure-free | 2 | 0 | 7
  Not seizure-free | 174 | 179 | 168

11. Secondary Outcome: Number of Participants Who Were Seizure-free During the Maintenance Phase
Description: Participants were considered to be seizure-free if they had not reported any seizures during the Maintenance Phase.
Time Frame: Week 5 through Week 16
Population: ITT EMEA Population
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 164 | 158 | 149
participants
  Seizure-free | 2 | 5 | 7
  Not seizure-free | 162 | 153 | 142

12. Secondary Outcome: Percentage of Seizure-free Days During the DB Phase (Titration and Maintenance Phases)
Description: A seizure-free day was a day without any seizures. For a participant to be seizure free during the DB Phase, the participant had to be seizure free both Week 7 to Week 18 and Week 1 to Week 6. A participant could be seizure free Week 7 to Week 18 (during the Maintenance Phase), but not seizure free Week 1 to Week 6. Hence, there are fewer participants being reported as seizure free from Week 1 to Week 18 than from Week 7 to Week 18. The percentage of seizure-free days was calculated as the total number of days without seizures in the DB period divided by the number of days in DB period x 100%.
Time Frame: Week 1 through Week 16
Population: ITT FDA Population. Only participants who had post-baseline seizure data were included in the analysis.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 176 | 179 | 175
percentage of days | 77.8 [0 to 100] | 79.5 [0 to 99] | 82.1 [0 to 100]

13. Secondary Outcome: Percentage of Seizure-free Days During the Maintenance Phase
Description: A seizure-free day was a day without any seizures. The percentage of seizure-free days was calculated as the total number of days without seizures in the Maintenance Phase divided by the number of days in the Maintenance Phase x 100%.
Time Frame: Week 5 through Week 16
Population: ITT EMEA Population
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 164 | 158 | 149
percentage of days | 78.1 [0 to 100] | 81.6 [0 to 100] | 84.5 [0 to 100]

14. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score at the End of the Maintenance Phase
Description: Clinical Global Impression of Improvement (CGI-I) is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the treatment. Scores on the scale are rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Week 16/end of treatment phase
Population: ITT EMEA Population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 164 | 158 | 149
scores on a scale | 3.2 (0.99) | 2.9 (1.05) | 2.9 (1.21)

15. Secondary Outcome: Patient Global Impression (PGI) Score at the End of the Maintenance Phase
Description: PGI is a participant-rated scale of improvement that was administered at the end of the Maintenance Phase in order to assess the participant's impression of his or her own improvement. PGI assessments were scored using a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Week 16/end of treatment phase
Population: ITT EMEA Population. Only participants with post-baseline PGI scores were included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 155 | 149 | 139
scores on a scale | 3.3 (1.00) | 2.9 (1.11) | 3.0 (1.43)

16. Secondary Outcome: Quality of Life Assessed by Quality of Life in Epilepsy-Problems Questionnaire (QOLIE-31-P) at BL (Week 0) and Weeks 4, 8, and 16
Description: The QOLIE-31-P is a 31-item questionnaire evaluating a participant's QOL perception in 7 domains: seizure worry, emotional well being, energy/fatigue, cognitive functioning, medication effects, social functioning, overall QOL. Precoded numeric values for some domains are such that a higher number reflects a more favorable health state; others are such that a higher number reflects a less favorable state. Precoded values are first converted to 0-100 point scores; higher converted scores always reflect better QOL. The overall score is derived by weighting and then summing the 7 domain scores.
Time Frame: End of Baseline (Week 0), Weeks 4, 8, and 16
Population: Safety Population: all randomized participants who received at least 1 dose of retigabine or placebo. Only participants with QOLIE-31-P data were included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 165 | 173 | 166
scores on a scale
  Baseline, n=165, 173, 166 | 53.3 (16.62) | 56.0 (17.45) | 52.1 (15.93)
  Week 4 (Titration Phase), n=155, 155, 149) | 55.4 (16.41) | 57.3 (18.12) | 52.7 (16.94)
  Week 8 (Maintenance Phase), n=141, 146, 127 | 55.3 (17.05) | 59.6 (17.32) | 52.7 (16.47)
  Week 16 (Maintenance Phase), n=143, 133, 123 | 54.7 (16.82) | 59.1 (16.57) | 53.2 (16.38)

17. Secondary Outcome: Number of Participants Whose Clinical Laboratory Values Were Deemed an Adverse Event by the Investigator (>=2% in Any Treatment Arm)
Description: Clinically important changes in laboratory values were to be reported as an adverse event if they met one of the following criteria: (1) intervention required; (2) change in dose of study drug required; (3) other treatment/therapy required; (4) association with other diagnoses.
Time Frame: Week 1 through Week 16
Population: Safety Population
Measure: Number; unit: participants
Groups:
- Placebo - Transition Phase: Participants receiving placebo during the Maintenance Phase were titrated to a target dose of retigabine 300 mg TID during the 4-week Transition Phase in a double-dummy, double-blind manner using a transition kit consisting of retigabine and placebo tablets (50 mg and 100 mg). The starting dose for retigabine titration was 100 mg TID and was increased weekly by a maximum of 150 mg per day
- Retigabine 200 mg TID - Transition Phase: Participants receiving retigabine 200 mg TID during the Maintenance Phase were titrated to a target dose of 300 mg TID retigabine during the 4-week Transition Phase in a double-dummy, double-blind manner using a transition kit consisting of retigabine and placebo tablets (50 mg and 100 mg). Retigabine doses were increased weekly by a maximum of 150 mg per day
- Retigabine 300 mg TID - Transition Phase: Participants receiving retigabine 300 mg TID during the Maintenance Phase continued receiving retigabine 300 mg TID during the 4-week Transition Phase in a double-dummy, double-blind manner using a transition kit consisting of retigabine and placebo tablets (50 mg and 100 mg). Placebo doses were administered to maintain the blinding and were increased weekly by a maximum of 150 mg per day
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance) | Placebo - Transition Phase | Retigabine 200 mg TID - Transition Phase | Retigabine 300 mg TID - Transition Phase
Number analyzed (Participants) | 179 | 181 | 178 | 147 | 132 | 114
participants
  Protenuria | 3 | 2 | 0 | 0 | 1 | 0
  Hyperlipidemia | 3 | 0 | 0 | 0 | 0 | 0
  Hypercholesterolemia | 2 | 4 | 1 | 0 | 0 | 1
  Hematuria | 2 | 5 | 2 | 1 | 0 | 1

18. Secondary Outcome: Number of Participants Who Reported the Indicated Renal and Urinary Disorder Adverse Events at a Frequency Threshold of 2% (in Any Treatment Arm)
Description: A summary of the adverse events classified as renal or urinary disorders and in which at least 2% (rounded to an integer) of participants in any treatment arm reported during the study is presented.
Time Frame: Week 1 through Week 16
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance) | Placebo - Transition Phase | Retigabine 200 mg TID - Transition Phase | Retigabine 300 mg TID - Transition Phase
Number analyzed (Participants) | 179 | 181 | 178 | 147 | 132 | 114
participants
  Dysuria | 0 | 3 | 4 | 0 | 0 | 0
  Urinary retention | 0 | 1 | 4 | 0 | 0 | 0
  Polyuria | 4 | 1 | 2 | 0 | 0 | 0
  Urinary hesitation | 3 | 6 | 1 | 3 | 1 | 0
  Haematuria | 2 | 5 | 2 | 1 | 0 | 1

19. Secondary Outcome: Change From Baseline in Post-void Residual Urine Volume at Weeks 8 and 16 of the Maintenance Phase
Description: Post-void residual (PVR) urine refers to the amount of urine remaining in the bladder after normal urination. To investigate the possible effects of retigabine on bladder function, all participants underwent post-void residual bladder ultrasound at Baseline and during the Maintenance Phase. The PVR bladder ultrasound was performed by a urologist, a qualified ultrasound technician, or a qualified study nurse who was certified to do PVR bladder ultrasound. Change from Baseline in PVR residual volume was calculated as the values at Week 10 and Week 16 minus the value at Baseline.
Time Frame: Baseline (Week -7 through 0), Weeks 8 and 16
Population: Safety Population. Only participants who remained in the study at the indicated week and who also had a PVR assessment were analyzed.
Measure: Median (Full Range); unit: milliliters
Groups:
- Placebo: Maintenance Phase: Matching placebo tablets of dummy strengths of 50 mg and 100 mg were administered orally TID during the 12-week Maintenance Phase
- Retigabine 200 mg TID: Maintenance Phase: Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 200 mg TID during the 12-week Maintenance Phase
- Retigabine 300 mg TID: Maintenance Phase: Retigabine 50 mg and 100 mg tablets were administered orally for a target dose of 300 mg TID during the 12-week Maintenance Phase
Arm/Group | Placebo: Maintenance Phase | Retigabine 200 mg TID: Maintenance Phase | Retigabine 300 mg TID: Maintenance Phase
Number analyzed (Participants) | 143 | 134 | 115
milliliters
  Week 8, n=143, 134, 121 | 0 [-107 to 148] | 0 [-195 to 400] | 0 [-162 to 165]
  Week 16, n=141, 131, 115 | 0 [-185 to 232] | 0 [-195 to 609] | 0 [-262 to 173]

20. Secondary Outcome: Number of Participants With a >=7% Increase in Body Weight During Weeks 2 and 4 of theTitration Phase and Weeks 6, 8, 12, and 16 of the Maintenance Phase
Description: The number of participants with recorded weight gain of >=7% over their baseline weight was measured.
Time Frame: Weeks 2 and 4 of Titration Phase and Weeks 6, 8, 12, and 16 of Maintenance Phase
Population: Safety Population. Only participants who remained in the study at the indicated week and who also had a body weight assessment were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance)
Number analyzed (Participants) | 174 | 180 | 175
participants
  Week 2, n=174, 180, 175 | 0 | 3 | 3
  Week 4, n=169, 172, 167 | 0 | 7 | 8
  Week 6, n=169, 165, 152 | 1 | 8 | 7
  Week 8, n=161, 160, 149 | 1 | 9 | 7
  Week 12, n=159, 151, 144 | 6 | 15 | 13
  Week 16, n=153, 139, 132 | 4 | 13 | 12

ADVERSE EVENTS:
Arm/Group | Placebo - Double Blind (DB) Phase (Titration Plus Maintenance) | Placebo - Transition Phase | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 200 mg TID - Transition Phase | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance) | Retigabine 300 mg TID - Transition Phase
Serious Adverse Events (participants affected / at risk) | 7/179 | 2/147 | 14/181 | 3/132 | 15/178 | 3/114
Other Adverse Events (participants affected / at risk) | 56/179 | 38/147 | 92/181 | 18/132 | 117/178 | 29/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Double Blind (DB) Phase (Titration Plus Maintenance) (N=179) | Placebo - Transition Phase (N=147) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) (N=181) | Retigabine 200 mg TID - Transition Phase (N=132) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance) (N=178) | Retigabine 300 mg TID - Transition Phase (N=114)
Convulsion (Nervous system disorders) | 1 | 0 | 3 | 2 | 3 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nerve root compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atonic urinary bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sudden unexplained death in epilepsy (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deja vu (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Corneal erosion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Visual disturbance (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Double Blind (DB) Phase (Titration Plus Maintenance) (N=179) | Placebo - Transition Phase (N=147) | Retigabine 200 mg TID - DB Phase (Titration Plus Maintenance) (N=181) | Retigabine 200 mg TID - Transition Phase (N=132) | Retigabine 300 mg TID - DB Phase (Titration Plus Maintenance) (N=178) | Retigabine 300 mg TID - Transition Phase (N=114)
Dizziness (Nervous system disorders) | 12 | 16 | 31 | 3 | 46 | 10
Somnolence (Nervous system disorders) | 18 | 9 | 26 | 3 | 46 | 12
Headache (Nervous system disorders) | 26 | 8 | 20 | 4 | 31 | 7
Fatigue (General disorders) | 5 | 2 | 30 | 2 | 27 | 2
Tremor (Nervous system disorders) | 4 | 2 | 3 | 1 | 16 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 1 | 15 | 1 | 12 | 2
Nausea (Gastrointestinal disorders) | 7 | 2 | 11 | 3 | 12 | 2
Asthenia (General disorders) | 4 | 2 | 9 | 2 | 12 | 4
Memory impairment (Nervous system disorders) | 3 | 2 | 7 | 1 | 11 | 1
Diplopia (Eye disorders) | 2 | 1 | 12 | 3 | 10 | 0
Disturbance in attention (Nervous system disorders) | 4 | 2 | 13 | 1 | 10 | 2
Vision blurred (Eye disorders) | 3 | 2 | 1 | 1 | 9 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 3 | 1 | 9 | 0
Coordination abnormal (Nervous system disorders) | 3 | 3 | 11 | 1 | 8 | 3
Gait disturbance (General disorders) | 1 | 1 | 6 | 0 | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.